CLINICAL TRIAL: NCT02023918
Title: Role of Growth Hormone Antagonism in Modulating Insulin Sensitivity in Subjects With Insulin Resistance But Without Diabetes
Brief Title: Role of Growth Hormone Antagonism in Modulating Insulin Sensitivity in Subjects With Pre-diabetes
Acronym: PEGIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI178028
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Metabolic Syndrome; Insulin Resistance
Keywords: Growth hormone antagonism
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Insulin Resistance | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegvisomant arm (Experimental): Pegvisomant 20 mg subcutaneously Qday x 28 days will be administered by the study subject.
  Interventions: Drug: pegvisomant

INTERVENTIONS:
Drug: pegvisomant — Pegvisomant 20 mg subcutaneously Qday will be administered by the study subject for 28 days during this study.
  Other Names: Somavert

SUMMARY:
Growth hormone is well known to cause changes in glucose regulation. People with Laron syndrome are born without the growth hormone receptor and are protected from diabetes. Mice who are engineered without the growth hormone receptor are similarly protected from diabetes. Conversely, people who have excessive amounts of growth hormone, such as patients with acromegaly, have an increased risk for type 2 diabetes. In acromegaly patients, treatment with pegvisomant, a medication that reduces insulin like growth factor-1 by blocking the growth hormone receptor, significantly improves insulin resistance. Pegvisomant has not been explored as a possibility for the treatment of type 2 diabetes or insulin resistance in people without acromegaly. In this study, the investigators hope to study the metabolic effects of pegvisomant on people who have insulin resistance but not diabetes. Pegivosmant is expected to improve insulin resistance in the liver, fat and muscle as well as decrease serum free fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-35
* Homeostatic model assessment - insulin resistance (HOMA-IR) >2.77
* Able to administer daily subcutaneous injections of pegvisomant

Exclusion Criteria:

* Pregnancy
* Breastfeeding in the last 6 months
* Liver function tests greater than 3x the upper limits of normal
* unstable diet over the last 3 months
* unstable weight over the last 6 months
* unstable lipid lowering regimen
* diabetes - type 1 or type 2
* History of major gastrointestinal surgery
* History of pancreatic, liver, biliary, or intestinal disease
* Fasting blood glucose >126
* Fasting triglycerides>500
* A1c>6.5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan J Weiss, MD, Principal Investigator — University of California, San Francisco; Morris Schambelan, MD, Principal Investigator — University of California, San Francisco; Kathleen Mulligan, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegvisomant Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pegvisomant Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Investigators will measure insulin sensitivity via hyperinsulinemic euglycemic clamp prior to the initiation of the study medication and then again at the end of the 28 days to evaluate the effect of pegvisomant on insulin sensitivity and reported as HOMA-IR.
  HOMA-IR was derived from fasting insulin and fasting glucose by the calculation: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5
Time Frame: 28 days
Population: Patients were compared after treatment to their own baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pegvisomant Arm
Number analyzed (Participants) | 6
units on a scale
  Baseline HOMA-IR | 3.06 (1.46)
  HOMA-IR after 28 days of treatment | 3.33 (2.76)

2. Secondary Outcome: Lipolysis
Description: Treatment with pegvisomant is expected to alter lipolysis. To assess this investigators will do fasting and steady state stable isotope measurements prior to treatment with pegvisomant and at day 28 after treatment with pegvisomant.
Time Frame: 28 days
Population: Ra glycerol reported
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Pegvisomant Arm
Number analyzed (Participants) | 6
mg/kg/min
  Ra glycerol fasting state baseline | 0.20 (0.07)
  Ra glycerol fasting state after 28 days of peg | 0.21 (0.02)
  Ra glycerol steady state baseline | -0.01 (0.2)
  Ra glycerol steady state treatment 28 days peg | 0.4 (0.2)

ADVERSE EVENTS:
Arm/Group | Pegvisomant Arm
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No